CLINICAL TRIAL: NCT01671774
Title: Multicenter, Open-label, Exploratory Phase I Pilot Study to Investigate Safety, Pharmacodynamics, and Pharmacokinetics of Immunological Effects and Activity of Combining Multiple Doses of IMAB362 With Immunomodulation (Zoledronic Acid, Interleukin-2) in Patients With Advanced Adenocarcinoma of the Stomach, the Lower Esophagus, or the Gastroesophageal Junction
Brief Title: Safety and Activity of IMAB362 in Combination With Zoledronic Acid and Interleukin-2 in CLDN18.2-positive Gastric Cancer
Acronym: PILOT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: GM-IMAB-001-04; 2011-005509-64 (EudraCT Number)
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: CLDN18.2-positive Gastric Adenocarcinoma; CLDN18.2-positive Adenocarcinoma of the Gastroesophageal Junction; CLDN18.2-positive Adenocarcinoma of Esophagus
MeSH Terms: interventions — zolbetuximab; Zoledronic Acid; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IMAB362 + ZA (Experimental): Participants received IMAB362 on Day 1 of each 3-week cycle (every 3 weeks). Participants received ZA on Day 1.
  Interventions: Drug: IMAB362; Drug: Zoledronic acid
- IMAB362 + ZA + IL-2 (1 million IU) (Experimental): Participants received IMAB362 on Day 1 of each 3-week cycle (every 3 weeks). Participants received ZA on Day 1 and IL-2 on Days 1 to 3 of Cycles 1 and 3 only.
  Interventions: Drug: IMAB362; Drug: Zoledronic acid; Drug: Interleukin-2 (1 million IU)
- IMAB362 + ZA + IL-2 (3 million IU) (Experimental): Participants received IMAB362 on Day 1 of each 3-week cycle (every 3 weeks). Participants received ZA on Day 1 and IL-2 on Days 1 to 3 of Cycles 1 and 3 only.
  Interventions: Drug: IMAB362; Drug: Zoledronic acid; Drug: Interleukin-2 (3 million IU)
- IMAB362 (Active Comparator): Participants received IMAB362 only on Day 1 of each cycle every 3 weeks.
  Interventions: Drug: IMAB362

INTERVENTIONS:
Drug: IMAB362 — 800 mg/m2 on d 1 of cycle 1. 600 mg/m2 on d 1 of every other cycle
Drug: Zoledronic acid — 4 mg on d 1 of cycle 1 and cycle 3
  Arms: IMAB362 + ZA; IMAB362 + ZA + IL-2 (1 million IU); IMAB362 + ZA + IL-2 (3 million IU)
Drug: Interleukin-2 (1 million IU) — 1 million IU on day 1, 2 and 3 of cycles 1 and 3.
  Arms: IMAB362 + ZA + IL-2 (1 million IU)
Drug: Interleukin-2 (3 million IU) — 3 million IU on day 1, 2 and 3 of cycles 1 and 3.
  Arms: IMAB362 + ZA + IL-2 (3 million IU)

SUMMARY:
The purpose of the trial is to assess the immunological effects and their kinetics, the safety and activity of IMAB362 plus Zoledronic acid with/without low to intermediate doses of Interleukin-2 in subjects with advanced gastroesophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach, the esophagus or the gastroesophageal junction
* Inoperable locally advanced disease, resections with R0, R1 or R2 outcome or metastatic disease.
* CLDN18.2 expression confirmed by immunohistochemistry in paraffin embedded tumor tissue sample.
* Measurable and/or non-measurable disease as defined according to RECIST v1.1
* Age ≥ 18 years
* Written informed consent
* ECOG performance status (PS) 0-1
* Life expectancy > 3 months

Exclusion Criteria:

* Prior hypersensitivity reaction or intolerance to one of the compounds of the study treatment
* Known HIV infection or known symptomatic hepatitis (A, B, C)
* Clinical symptoms of cerebral metastases
* Pregnancy or breastfeeding
* Patients treated with any bisphosphonate-based therapeutic for any indication during the previous year
* Hypocalcemia that requires medication. Corrected (adjusted for serum albumin) serum calcium < 8 mg/dl (2 mmol/L) or > 12 mg/dL (3.0 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2014-10-13 (Actual); Study Completion 2014-10-13 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | at least 18 months
  Descriptive statistics for treatments will be given on the number of patients whose treatment had to be reduced, delayed or permanently stopped.
Immune cell profile and kinetics | at least 18 months
  Descriptive statistics for treatments will be given on the number and activity of immune cells in peripheral blood of patients.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | at least 18 months
  PFS is defined as the time from registration of therapy to the first observation of disease progression or death from any cause or last tumor evaluation if free of progression. For patients who have not progressed either clinically or on the last scan, they will be censured as of the last tumor evaluation.
Objective tumor response rate (ORR) | at least 18 months
  ORR comprises the fraction of patients with CR, PR according to RECIST v1.1. It is set in relation to the ITT population and PP population.
Disease control rate (DCR) | at least 18 months
  DCR is defined as the fraction of patients with CR or PR or SD according to RECIST v1.1. It is set in relation to the ITT population and PP population.
Duration of response (DOR) | at least 18 months
  Duration of response is determined as the time when criteria for CR, PR, and SD are first met until the first date that recurrent or progressive disease or death occurs.

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (7):
  - Institut für Klinische Forschung, Krankenhaus Nordwest GmbH, Frankfurt am Main, Hesse
  - BAG / Onkologische Schwerpunktpraxis, Dresden, Saxony
  - Charité Universitätsmedizin Berlin - CVK, Med. Klinik m.S. Hämatologie und Onkologie, Berlin
  - Freiburg University Medical Center, Department of Internal Medicine II, Gastroenterology and Hepatology, Freiburg im Breisgau
  - Leipzig University Hospital, University Cancer Center (UCCL), Leipzig
  - University Hospital Tuebingen, Department of Internal Medicine I - Gastroenterology, Hepatology, Infectious Diseases, Tübingen
  - Ulm University Hospital, Center for Internal Medicine, Ulm
- Latvia (2):
  - Piejuras Hospital, Oncology Clinic, Liepāja
  - Riga East University Hospital, LLC, Latvian Oncology Center, Riga

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Lordick F, Thuss-Patience P, Bitzer M, Maurus D, Sahin U, Tureci O. Immunological effects and activity of multiple doses of zolbetuximab in combination with zoledronic acid and interleukin-2 in a phase 1 study in patients with advanced gastric and gastroesophageal junction cancer. J Cancer Res Clin Oncol. 2023 Aug;149(9):5937-5950. doi: 10.1007/s00432-022-04459-3. Epub 2023 Jan 6. PMID 36607429
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=25767&tenant=MT_AST_9011